CLINICAL TRIAL: NCT04211103
Title: Single Arm Phase II Study on Pembrolizumab in Pre Neoplastic High Grade HPV-related Vulvar and Cervical Lesions
Brief Title: Pembrolizumab in Pre Neoplastic High Grade HPV-related Vulvar and Cervical Lesions
Acronym: MITO CERV 4
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2773
Record Dates: First submitted 2019-12-22; First posted 2019-12-26 (Actual); Last update posted 2021-08-27 (Actual); Status verified 2021-08

CONDITIONS: Cervical, Vaginal and Vulval Inflammatory Diseases
MeSH Terms: interventions — pembrolizumab

STUDY DESIGN:
Intervention Model Description: single arm phase II trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pembrolizumab single agent (Experimental): Pembrolizumab single agent as neoadjuvant treatment before surgical conization and/or partial or radical vulvectomy.
  Pembrolizumab 200 mg flat dose will be administered every 3 weeks for 5 cycles. Within 3 weeks from the last Pembrolizumab administration patients will be submitted to surgical conization or partial or radical vulvectomy.
  Interventions: Drug: Pembrolizumab

INTERVENTIONS:
Drug: Pembrolizumab — Humanized antibody used in cancer immunotherapy. It targets the programmed cell death protein 1 (PD-1) receptor of lymphocytes.
  Other Names: Keytruda

SUMMARY:
single arm phase II trial evaluating Pembrolizumab single agent as neoadjuvant treatment before surgical conization and/or partial or radical vulvectomy in patients with pre-neoplastic cervical and vulvar high grade lesions.

DETAILED DESCRIPTION:
This is a single arm phase II trial evaluating Pembrolizumab single agent as neoadjuvant treatment before surgical conization and/or partial or radical vulvectomy in patients with pre-neoplastic cervical and vulvar high grade lesions. Patients with histologically confirmed H-SIL and/or VIN 2-3 lesions will be treated with Pembrolizumab 200 mg flat dose every 3 weeks for 5 cycles. Within 3 weeks from the last Pembrolizumab administration patients will be submitted to surgical conization or partial or radical vulvectomy.

ELIGIBILITY:
Inclusion Criteria:

1. Female participants who are at least 18 years of age on the day of signing informed consent with histologically confirmed diagnosis of cervical HSIL OR vulvar VIN 2-3 lesions will be enrolled in this study.
2. A female participant is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies:

   1. Not a woman of childbearing potential (WOCBP) OR
   2. A WOCBP who agrees to follow the contraceptive guidance during the treatment period and for at least 3 months after the last dose of study treatment.
3. The participant (or legally acceptable representative if applicable) provides written informed consent for the trial.
4. Have provided archival tumor tissue sample (if pre treatment biopsy performed at other institution) or newly obtained core or excisional biopsy of the lesion. Formalin-fixed, paraffin embedded (FFPE) tissue blocks are preferred to slides. Newly obtained biopsies are preferred to archived tissue.

   Note: If submitting unstained cut slides, newly cut slides should be submitted to the testing laboratory within 14 days from the date slides are cut.
5. Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1. Evaluation of ECOG is to be performed within 7 days prior to the date of registration .
6. Have adequate organ function as defined in the following table (Table 1). Specimens must be collected within 10 days prior to the start of study treatment.

Exclusion Criteria:

1. A WOCBP who has a positive urine pregnancy test within 72 hours prior to study drug treatment. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.

   Note: in the event that 72 hours have elapsed between the screening pregnancy test and the first dose of study treatment, another pregnancy test (urine or serum) must be performed and must be negative in order for subject to start receiving study medication.
2. Has received prior therapy with an anti-PD-1, anti-PD-L1, or antiPDL2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (eg, CTLA-4, OX40, CD137).
3. Has received prior systemic anti-cancer therapy including investigational agents within 4 weeks [could consider shorter interval for kinase inhibitors or other short half-life drugs] prior to [randomization /allocation].

   Note: Participants must have recovered from all AEs due to previous therapies to ≤Grade 1 or baseline. Participants with ≤Grade 2 neuropathy may be eligible.

   Note: If participant received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting study treatment.
4. Has received prior radiotherapy within 2 weeks of start of study treatment. Participants must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis. A 1-week washout is permitted for palliative radiation (≤2 weeks of radiotherapy) to non-CNS disease.
5. Has received a live vaccine within 30 days prior to the first dose of study drug. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guérin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (eg, FluMist®) are live attenuated vaccines and are not allowed.
6. Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study treatment.

   Note: Participants who have entered the follow-up phase of an investigational study may participate as long as it has been 4 weeks after the last dose of the previous investigational agent.
7. Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug.
8. Has a known additional malignancy that is progressing or has required active treatment within the past 3 years. Note: Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ (e.g. breast carcinoma) that have undergone potentially curative therapy are not excluded.
9. Has known active CNS metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate provided they are radiologically stable, i.e. without evidence of progression for at least 4 weeks by repeat imaging (note that the repeat imaging should be performed during study screening), clinically stable and without requirement of steroid treatment for at least 14 days prior to first dose of study treatment.
10. Has severe hypersensitivity (≥Grade 3) to pembrolizumab and/or any of its excipients.
11. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
12. Has a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis.
13. Has an active infection requiring systemic therapy.
14. Has a known history of Human Immunodeficiency Virus (HIV). Note: No HIV testing is required unless mandated by local health authority.
15. Has a known history of Hepatitis B (defined as Hepatitis B surface antigen [HBsAg] reactive) or known active Hepatitis C virus (defined as qualitative HCV RNA is detected) infection. Note: no testing for Hepatitis B and Hepatitis C is required unless mandated by local health authority.
16. Has a known history of active TB (Bacillus Tuberculosis).
17. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
18. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
19. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of trial treatment.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2020-10-14 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Efficacy of Pembrolizumab: proportion of subjects with no evidence of cervical HSIL on histology at surgical treatment | 18 months
  proportion of subjects with no evidence of cervical HSIL on histology at surgical treatment

SECONDARY OUTCOMES:
Efficacy of Pembrolizumab: Proportion of subjects with no evidence of vulvar VIN 2-3 on histology at surgical treatment | 18 months
  Proportion of subjects with no evidence of vulvar VIN 2-3 on histology at surgical treatment
Efficacy of Pembrolizumab: Incidence and severity of systemic events for the duration of the study (CTCAE 5.0) | 18 months
  Incidence and severity of systemic events for the duration of the study (CTCAE 5.0)
Efficacy of Pembrolizumab: Proportion of subjects with downstaging of cervical and vulvar pre-neoplastic lesion on histology | 18 months
  Proportion of subjects with downstaging of cervical and vulvar pre-neoplastic lesion on histology
Efficacy of Pembrolizumab: Proportion of patients with no evidence of HPV by HPV testing at Week 36 visit | 18 months
  Proportion of patients with no evidence of HPV by HPV testing at Week 36 visit
Efficacy of Pembrolizumab: Proportion of subjects with no progression of cervical HSIL and vulvar VIN 2-3 to cervical and vulvar carcinoma respectively from baseline on histology | 18 months
  Proportion of subjects with no progression of cervical HSIL and vulvar VIN 2-3 to cervical and vulvar carcinoma respectively from baseline on histology

CONTACTS AND LOCATIONS:
Locations (9):
- Italy (9):
  - Centro di Riferimento Oncologico, Aviano
  - Policlinico S.Orsola-Malpighi, Bologna
  - Ospedale "degli Infermi", Faenza
  - Ospedale "Umberto I", Lugo
  - Ospedale Sacro Cuore Don Calabria, Negrar
  - Ospedale Santa Maria delle Croci, Ravenna
  - Ospedale Infermi, Rimini
  - Fondazione Policlinico Universitario A. Gemelli IRCCS, Rome
  - Istituti fisioterapici Ospitalieri - Istituto Tumori Regina Elena, Rome

IPD SHARING:
Plan to Share IPD: No